CLINICAL TRIAL: NCT05293119
Title: Efficacy of Tofacitinib in Vitiligo-a Randomized Controlled Trial in a Selected Tertiary Level Hospital in Dhaka
Brief Title: Role of Tofacitinib in Vitiligo Patients
Acronym: ETV
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pi Research Consultancy Center, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pircc-1026
Record Dates: First submitted 2021-06-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Vitiligo; Effect of Drug
Keywords: Vitiligo; Tofacitinib; Dermatology; Skin
MeSH Terms: conditions — Vitiligo | interventions — tofacitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: The participants will undergo randomization into 1:1 ratio into two equal groups. Group A will receive oral Tofacitinib and Group B will receive topical 0.1%Mometasone furoate. All the participants will receive allotted intervention for 12weeks. The patient will be followed up at 6 weeks and end of 12 weeks. Primary outcome of the study will be improvement of Vitiligo Area Scoring Index (VASI) score at 6 and12 weeks in all groups. Secondary outcomes will include improvement in Vitiligo European Task Force (VETF) scoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tofacitinib (Experimental): In this group, study participants will be treated with per oral tofacitinib citrate (5 mg/twice daily)
  Interventions: Drug: JAK-2 inhibitor
- Topical corticosteroid (Active Comparator): In this group, patients will apply topical Mometasone furoate 0.1% once daily
  Interventions: Drug: Topical corticosteroid

INTERVENTIONS:
Drug: JAK-2 inhibitor — In this trial, one group will receive the tofacitinib 5 mg twice daily
  Other Names: Tofacitinib
  Arms: Tofacitinib
Drug: Topical corticosteroid — Mometasone furoate 0.1% ointment once daily
  Other Names: Mometasone furoate 0.1%
  Arms: Topical corticosteroid

SUMMARY:
Standard treatment for vitiligo often has unsatisfactory outcomes. With a new understanding of pathogenesis, novel drugs have been introduced which have shown to be effective in small-scale studies. Tofacitinib, a Janus kinase(JAK) inhibitor-2 has shown promising results in the treatment of vitiligo. However, randomized controlled studies are required to confirm these observations and identify the patients most likely to benefit from JAK-2 inhibition. This open-labeled randomized clinical trial will be conducted at the department of dermatology and venereology of US Bangla Medical College & Hospital in Dhaka for 6 months duration from June 2021 to November 2021 to Vitiligo patients attending in the aforementioned department will be approached for inclusion in the study. Finally, 80 patients who will fulfill the inclusion and exclusion criteria will be included. All patients will be informed about the nature of the study and the written consent will be taken in the consent form with the assurance that their information will be made confidential. Baseline information such as gender, age, disease history, and drugs used prior will be collected. All patients will undergo baseline laboratory evaluation which will be repeated at 6weeks and 12weeks. Before the beginning of treatment, digital images of the cutaneous lesions will be taken which will be compared with the ones taken at 6weeks and the end of 12weeks follow up. The participants will undergo randomization into 1:1 ratio into two equal groups. Group A will receive oral Tofacitinib and Group B will receive topical 0.1%Mometasone furoate. All the participants will receive allotted intervention for 12weeks. The patient will be followed up at 6 weeks and end of 12 weeks. The primary outcome of the study will be the improvement of the Vitiligo Area Scoring Index (VASI) score at 6 and12 weeks in all groups. Secondary outcomes will include improvement in Vitiligo European Task Force (VETF) scoring. The data will be systematically described and summarized and presented through descriptive statistics and finally will be analyzed by the statistical program Statistical Package for Social Science (SPSS) version 23.0(Chicago, Illinois, USA). The relevant statistical test will be used during the analysis. In all cases, the significance level will set p <0.05. Ethical clearance of the study will be obtained from the ethical review committee (ERC) of the study place.

DETAILED DESCRIPTION:
Participant selection:

All vitiligo irrespective of the duration of the disease presenting at the outpatient department will be initially approached for inclusion in the study. Eighty patients who will fulfillthe inclusion criteria will be recruited inthe study. The patients will be briefed about the aim, objective and details of the procedure the study.

Consent & recruitment:

Participant information sheets will be provided for all trial participants, and ample opportunity is given to discuss the study with the investigator before agreeing to take part. All participants will provide written informed consent for participation, retention and use of the trial data by members of the research group (use of the trial photo-graphs for further research or trial reporting is optional).

Baseline information:

Clinical and demographic information, including sex, age, Fitzpatrick type of skin, disease duration and course, medical history, family history and prior treatment will be collected. Baseline laboratory testing (complete blood count, liver function tests, renal function test, basic metabolic panel, hepatitis B/C panel, Tuberculosis and HIV screening) will be performed.

Baseline Vitiligo Area Scoring Index (VASI) score:

Hamzavi et al.19 have introduced a quantitative parametric score, named VASI for Vitiligo Area Scoring Index. The total body VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100) Total Body surface area (BSA) will be calculated with the use of a handprint (palm plus the volar surface of fingertips) to estimate 1% BSA. Multiplication of affected BSA (estimated with the use of hand units) by the degree of depigmentation (0-100%) within each hand unit will be performed to calculate a VASI score.

Baseline Vitiligo European Task Force(VETF) scoring:

Baseline extent of disease, staging, and spread will be measured according to Vitiligo European Task Force scoring tool.

Digital images of the cutaneous lesions, both with normal ambient light and with Wood's lamp, will be obtained before the treatment beginning and at 6 weeks and 12 weeks(at the end of study).

Washout of previous treatment:

Patients with recent vitiligo treatment exposure will be required to wash out of treatment within designated time frames (topical treatment, 2 weeks; immunomodulating oral medications, 4 weeks; laser and light treatment, 8 weeks; and investigational/biologic therapies, 12 weeks). Patients will be asked to refrain from using other vitiligo treatments throughout the duration of the trial.

Confidentiality:

Trial data and individual participants' medical information obtained as a result of this study is considered confidential. Participant confidentiality will be ensured by using identification code numbers to correspond to treatment data in the computer files and on trial photographs.

Participant timeline Participants are enrolled in the trial for 6 months. During this period, participants attend a hospital outdoor at baseline for recruitment, medical photography, photo-sensitivity assessment (minimum erythema dose (MED) test) and followed by assessment at 6 and 12 weeks for compliance and outcome.

Randomization and blinding

Participants are randomized to one of two treatment groups in a ratio of 1:1 where each group has equal opportunity to receive any treatment option as follows:

Tofacitinib group (Group A) Topical corticosteroid group (Group B) After all eligibility criteria have been confirmed and medical photographs taken, participants are randomized by lottery. Participants, principal investigators, members of trial management group and data analysts are not blinded to treatment allocation.

Interventions:

Tofacitinib: (Group A) Treatment with oral tofacitinib citrate, will be initiated with, 5mg, twice daily. It is associated with infections, malignancies, cytopenias, gastrointestinal perforations and hyperlipidaemia in some patients with rheumatoid arthritis.

Topical corticosteroid: (Group B) Mometasone furoate 0.1% ointment a potent corticosteroid used once daily, has been recommended in the European Clinical Guidelines for the management of vitiligo. In order to minimize the risk of adverse reactions, the Guidelines recommend a discontinuous regimen involving periods of use followed by break periods. Possible adverse reactions to mometasone furoate 0.1% include: infection, folliculitis, paraesthesia, burning sensation, contact dermatitis, skin hypopigmentation, hypertrichosis, skin striae, acneiform dermatitis, skin atrophy, pruritus, application site pain and visual disturbance. Participants are advised to stop treatment with the ointment if they notice any side effects and to contact the local research team for review and advice on when to restart treatment.

Adherence:

Adherence is recorded in a treatment diary, which acts as a record to inform clinic appointment questions about the number of ointment applications undertaken since the last clinic visit. Collection of these data at each clinic visit (every 6weeks) also helps to check participants' understanding of treatment and to encourage adherence; additional training is provided at the clinic visit if it has been noticed the participant is not using the device appropriately or has misunderstood the treatment schedule.

Treatment modification following adverse events:

Participants are instructed to record adverse events in their treatment diaries and to contact their recruiting center if they experience side effects of concern, or a serious adverse event (whether related to the trial treatment or not). For treatment-related side effects, or drug-induced photosensitivity, the research team provides telephone advice or arrange for a dermatology consultation, as necessary. Treatment modifications, including reduction or suspension (temporary or permanent) of either oral tofacitinib, topical corticosteroid at the discretion of the dermatologist, as appropriate.

In case of a medical emergency where an active treatment of the oral drug or the device would need to be stopped, active treatment of both interventions should be assumed.

Data collection and management:

Data collection and skin assessments will be undertaken by the investigators at the recruiting hospital. Participants will be assessed end of6 weeks and 12 weeks with observation of improvement in regards to re-pigmentation, extent of disease, staging, and spread. Photographs of the lesion will be taken during each visit and the participants will be inquired and examined to find out side effects of the interventions. Participants who do not attend clinic visits at 6 weeks and 12 weeks continue to be invited to subsequent follow-up visits unless they decline further participation in the trial. Laboratory testing (complete blood count, liver function tests, renal function test, basic metabolic panel will be performed at 6 weeks and 12 weeks.

Outcomes:

Primary outcome:

The primary outcome will be improvement in the VASI 6 weeks and 12 weeks. Multiplication of affected BSA (estimated with the use of hand units) by the degree of depigmentation (0-100%) within each hand unit was performed to calculate a VASI score (possible range, 0-100).

Secondary outcome:

Secondary outcomes included improvement in Vitiligo European Task Force scoring. The Vitiligo European Task Force is a validated tool that grades vitiligo on extent of disease, staging, and spread. Extent of disease is calculated by use of the "rule of nine" to estimate BSA, staging is assessed through degree of depigmentation on a 0 (no depigmentation) to 4 (complete depigmentation) scale, and spread is scored on a simple scale (+1: progressive; 0: stable; -1: regressive).

Withdrawal of study participants:

Participants are free to withdraw from the study at any point, for any reason. If this occurs, the primary reason for withdrawal will be documented in the participant's case record form. The participant will have the option of withdrawal from:

* Study medication with continued study procedures and collection of clinical and safety data,
* All aspects of the trial but continued use of data collected up to that point
* All aspects of the trial with the removal of all previously collected data, or
* All aspects of the trial with the removal of previously collected data and stored participant samples Randomized patients who wish to withdraw from the study before they have undertaken any study-related procedures will be replaced. Data on the original participant will be kept on the case record form (CRF)/database if the participant agrees to this.

Storage:

Drugs will be stored at room temperature 20-250 in trial storage room. Reconstituted solution with Bacteriostatic water for injection will also be kept at temperature 20-250.

Prohibited Medications: Any interventions for vitiligo, beside those provided in the trial are specifically prohibited.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Vitiligo patients
* Willing to participate

Exclusion Criteria:

* Age <18 years
* Patients with leukoderma secondary to other causes
* Participants with segmental or universal vitiligo
* Rapidly spreading vitiligo
* Lesions on areas known to be recalcitrant to therapy such as mucosal vitiligo
* Participants with a history of skin cancer
* Radiotherapy use
* Photosensitivity
* Women who are pregnant, breastfeeding or likely to become pregnant during the 9-month treatment period;
* Those currently using immunosuppressive drugs
* Involved in another clinical trial
* Not willing to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the VASI at 6 weeks. | 6 weeks
  The primary outcome will be a change in the VASI score at 6 weeks
Change in the VASI at 12 weeks | 12 weeks
  The primary outcome will be a change in the VASI score at 12 weeks

SECONDARY OUTCOMES:
Change in Vitiligo at 6th week by Vitiligo European Task Force scoring | 6 weeks
  Secondary outcomes included a change in Vitiligo European Task Force scoring
Change in Vitiligo at 12th week by Vitiligo European Task Force scoring | 12 weeks
  Secondary outcomes included a change in Vitiligo European Task Force scoring

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jahid Hasan, MPH, Study Chair — Pi Research Consultancy Center, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Data entry will be done in coded way and anonymously, so there will be very little chance to breach the Confidentiality of the patients.